CLINICAL TRIAL: NCT03498742
Title: Asthmatic Subjects Could Live Without Short Acting Beta2 Agonists (SABA)
Brief Title: Asthmatic Subjects Could Live Without Short Acting beta2 Agonists
Acronym: NOSABA
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Principal Investigator, HEEP UNR, Pulmonologist in Chief Pulmonary Section HEEP, Universidad Nacional de Rosario
Other Study IDs: HEEP-UNR-No SABA-02
Record Dates: First submitted 2018-04-02; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Asthma Chronic
Keywords: asthma; SABA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No SABA users: Asthmatic subjects that did not use short acting beta2 agonists in the last 3 months and being using none agent or ICS, systemic corticosteroids of combined ICS/LABA as relief symptoms agent.
  Interventions: Other: NO Intervention
- SABA users: Most of the asthmatic subjects usually inhale SABA as rescue medication and many times SABA is the only one prescribed treatment for asthma.
  Interventions: Other: NO Intervention

INTERVENTIONS:
Other: NO Intervention — Routine clinical data; asthma control test and spirometry
  Other Names: Self-administered asthma control test and spirometry.

SUMMARY:
Since 2006 there was a plateau in world wide mortality from asthma. Overreliance in Short Acting Beta2 Agonists (SABA) was associated with increased risk of death from asthma. Long acting beta agonists (LABA) alone was not permitted as treatment for asthma as it was determined by FDA by the "black box". By contrast SABA does not have a "black box", despite similar overuse alerts associated with increased risk of death from asthma. the investigators want to know if exist asthmatic subjects that do use another rescue medication; not SABA, and to compare their features, Asthma Control Test (ACT), and lung function in a outpatient facility.

First consecutive visits at outpatient Pulmonary Section of asthmatic subjects were described. Asthma Control Test (ACT) that was routinely used to assess asthma and spirometry were performed.

DETAILED DESCRIPTION:
During the period from March 10, 2017 to January 16, 2018 the investigators decided to describe the rescue medication in all new asthmatic subjects that came for a first visit to the outpatient pulmonary department. Patients aged ≥16 years were entered in the study with a a diagnosis of asthma, based on a history of episodic dyspnea and wheezing, and/or documented bronchodilator reversibility in forced expiratory volume in 1 s (FEV1) of 12% and 200 ml according to the National Institutes of Health criteria; to be non- or ex-smoker of less than 10 pack-yr, to be neither pregnant nor breast-feeding and to be capable of completing Asthma control test and spirometry. Consecutive patients visiting the outpatient pulmonary department were included in the description.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of asthma, based on a history of episodic dyspnea and wheezing, and/or documented bronchodilator reversibility in forced expiratory volume in 1 s (FEV1) of 12% and 200 ml according to the National Institutes of Health criteria;
2. to be non- or ex-smoker of less than 10 pack-yr,
3. to be neither pregnant nor breast-feeding
4. to be capable of completing Asthma control test and spirometry. -

Exclusion Criteria:

Any other pulmonary disorder than asthma. Illiteracy.

-

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients coming for a first visit to the Pulmonary Section, not only due to asthma; but also for presurgical assessment and/or Spirometry prescription.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test | One year
  Score less than 16 indicates Poorly controlled asthma. Score >19 indicates well controlled asthma.

SECONDARY OUTCOMES:
Acute asthma attack requiring Hospitalization and/or Emergency Room visits in the last 12 months | One year
  Stay for more than 24 hs in the Emergency and/or Hospitalization due to acute asthma exacerbations in the 12 months before the current visit

CONTACTS AND LOCATIONS:
Overall Officials: Luis J Nannini, MD, Principal Investigator — Universidad Nacional de Rosario
Locations (1):
- Pulmonary Section, Granadero Baigorria, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Corresponding author (Luis J Nannini) shared all the available data of this observational not interventional study with the other 3 investigators.
Supporting Information: Study Protocol, CSR
Time Frame: From March 20 2018 until desired publication

REFERENCES:
- [Background] Nannini LJ, Neumayer NS. Treatment Step 1 for Asthma Should Not Be Left Blank, and SABA-Only Might Not Be a Treatment Step 1 Option for Asthma. Respiration. 2018;95(3):212-214. doi: 10.1159/000484568. Epub 2017 Dec 14. No abstract available. PMID 29241185
- [Background] Rodrigo GJ, Arcos JP, Nannini LJ, Neffen H, Broin MG, Contrera M, Pineyro L. Reliability and factor analysis of the Spanish version of the asthma control test. Ann Allergy Asthma Immunol. 2008 Jan;100(1):17-22. doi: 10.1016/S1081-1206(10)60399-7. PMID 18254477